CLINICAL TRIAL: NCT04156542
Title: Measuring the Long-Term Impact of Behavioral Interventions in Middle School Cafeterias
Brief Title: Nudging for Behavior Change in School Cafeterias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Cornell University (Other); Columbus City School District (Unknown)
Responsible Party: Principal Investigator, Andrew Hanks, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016B0004; 2019B0480 (Other: Ohio State University); 62140-10509 (Other Grant/Funding Number: Cornell University)
Record Dates: First submitted 2019-10-29; First posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Behavior, Child; Food Selection
Keywords: Behavioral nudges; Food environment; Choice architecture; Lasting behavior change; Child nutrition; National School Lunch Program
MeSH Terms: conditions — Child Behavior; Food Preferences

STUDY DESIGN:
Intervention Model Description: We randomly assigned the six participating schools to either be a control school (N=1) or a treatment school (N=5). Each of the treatment schools administered a single intervention, but at different times. In our fifteen-week study, one school implemented the intervention for five weeks after five weeks of baseline data collection. Once this school completed the five weeks with the treatment, it removed the intervention and collected five more weeks of post-intervention data. In the other four schools, we staggered intervention implementation. The first school implemented the intervention on the first day of the study. The next school implemented the intervention after three weeks of collecting baseline data. The next school implemented the intervention after six weeks of collecting baseline data. Lastly, the final school implemented the intervention after nine weeks of collecting baseline data.
Who Masked: Participant
Masking Description: Researchers entered school cafeterias to collect student tray waste data. When students asked why the researchers were there, researchers indicated their purpose was to learn more about the National School Lunch Program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control (No Intervention): In this school, we collected data throughout the entire study without implementing any intervention.
- 5-week Intervention with Post-intervention Data Collection (Experimental): In this school, we collected baseline data for 5 weeks, implemented the intervention for five weeks, then removed the intervention and collected post-intervention data for five weeks.
  Interventions: Behavioral: Basic School Lunchroom Nudges
- Implement intervention for 15 weeks (Experimental): In this school, we implemented the intervention on January 11, 2016, the day the study began.
  Interventions: Behavioral: Basic School Lunchroom Nudges
- Implement intervention for 12 weeks (Experimental): In this school, we collected baseline data for three weeks and then implemented the intervention for the remaining twelve weeks.
  Interventions: Behavioral: Basic School Lunchroom Nudges
- Implement intervention for 9 weeks (Experimental): In this school, we collected baseline data for six weeks and then implemented the intervention for the remaining nine weeks.
  Interventions: Behavioral: Basic School Lunchroom Nudges
- Implement intervention for 6 weeks (Experimental): In this school, we collected baseline data for nine weeks and then implemented the intervention for the remaining six weeks.
  Interventions: Behavioral: Basic School Lunchroom Nudges

INTERVENTIONS:
Behavioral: Basic School Lunchroom Nudges — The intervention consists of three components: 1) serving fresh fruit in attractive bowls in at least two locations on the lunch line; 2) providing descriptive names for the vegetables; and 3) increasing amount of plain milk availability by 10% and placing it in front of the chocolate milk. For the vegetable naming intervention, researchers first developed, printed, and laminated descriptive vegetable name cards (2"x4"). Some examples included "Savory Collard Greens," and "[School Mascot] Salad." Cafeteria staff affixed name cards to the serving line sneeze-guards in front of the vegetables for the day. For the fruit intervention, we purchased and delivered two ceramic bowls to the intervention school. The cafeteria staff filled the bowls and put them in different locations on the lunch line. For the milk intervention, cafeteria staff increased the amount of plain milk available by 10% and placed plain in front of chocolate milk in the coolers.
  Arms: 5-week Intervention with Post-intervention Data Collection; Implement intervention for 12 weeks; Implement intervention for 15 weeks; Implement intervention for 6 weeks; Implement intervention for 9 weeks

SUMMARY:
The main purpose of this research is to look at a school lunchroom intervention that is known to improve fruit, vegetable, and milk consumption and see how it changes in the long run and if it affects the child's behavior permanently. The intervention will include the giving the vegetables descriptive names, moving the fruit to right next to the register and in attractive bowls, and increasing the amount of white milk served by 10%. The main forms of analyzing these results are through food preparation records, lunch sales records, and tray waste records. The first focus of this study is to see if there is a specific point in an intervention when improvement stops and therefore the intervention needs to be updated. This procedure involves looking at five similar middle schools with this same intervention over a 15 week period. The time of intervention implementation will vary by three week intervals, so the first will start the first week of school, the next school will start after three weeks of school, the next will start after six weeks of school, and the next will start after nine weeks of school, and the last will be a control school where there will be no intervention implementation. These intervals will help eliminate bias dealing with the beginning of the year excitement and seasonal effects. Food preparation records and lunch sales records will be collected from the school for the 15 week period. Tray waste will be recorded by having 200 randomly selected trays measured and collected twice a week over the 15 week period. This focus will help schools manage when they need to change their intervention so that improvements will not stop. The second focus of this study is to see if the children's improvement is kept when the intervention has stopped. This procedure will involve looking at a similar school to the other 5 schools. But unlike the other schools, this one will have the first 5 weeks without the intervention, then 5 weeks with the intervention, and then another 5 weeks without the intervention. Food preparation records and lunch sales records will be collected from the school for the 15 week period. Tray waste will be recorded by having 200 randomly selected trays measured and collected twice a week over the 15 week period. This second focus will help identify how effective this intervention is in permanently changing dietary habits.

ELIGIBILITY:
Inclusion Criteria:

* This research focused on food choices of middle school students, grades 6-8, which generally range in ages 11-14. In addition, since we are interested in learning about the types of cafeteria foods children select and what they throw away, we focus on students who receive a school lunch meal.

Exclusion Criteria:

* We exclude students who do not receive a school lunch meal.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3000 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2016-04-27 (Actual); Study Completion 2016-04-29 (Actual)

PRIMARY OUTCOMES:
Percentage of students that took a serving of fruit | 30 days
  To determine whether or not a student took a serving of fruit, we will rely on tray waste records that we collected twice a week (repeated measures) for the duration of the study. Based on these records, if a student selected a serving of fruit, she will receive a value of one. Otherwise, she will receive a value of zero. We will use this binary measure to estimate the proportion of students who took a serving of fruit.
Percentage of students that took a serving of vegetables | 30 days
  To determine whether or not a student took a serving of vegetables, we will rely on tray waste records that we collected twice a week (repeated measures) for the duration of the study. Based on these records, if a student selected a serving of vegetables, she will receive a value of one. Otherwise, she will receive a value of zero. We will use this binary measure to estimate the proportion of students who took a serving of vegetables.
Percentage of students that took a carton of white milk (one pint) | 30 days
  To determine whether or not a student took a carton of white milk, we will rely on tray waste records that we collected twice a week (repeated measures) for the duration of the study. Based on these records, if a student selected a carton of white milk, she will receive a value of one. Otherwise, she will receive a value of zero. We will use this binary measure to estimate the proportion of students who took a carton of white milk.
Percentage of students that took a serving of flavored milk (one pint) | 30 days
  To determine whether or not a student took a carton of flavored milk, we will rely on tray waste records that we collected twice a week (repeated measures) for the duration of the study. Based on these records, if a student selected a carton of flavored milk, she will receive a value of one. Otherwise, she will receive a value of zero. We will use this binary measure to estimate the proportion of students who took a carton of flavored milk.
Percentage of students that took an entree | 30 days
  To determine whether or not a student took an entree, we will rely on tray waste records that we collected twice a week (repeated measures) for the duration of the study. Based on these records, if a student selected an entree, she will receive a value of one. Otherwise, she will receive a value of zero. We will use this binary measure to estimate the proportion of students who took an entree.
Fraction of fruit serving wasted by the student | 30 days
  The tray waste records our researchers collected twice a week (repeated measures) for the duration of the study indicate how much -- 0, one-quarter, one-half, three-quarters, all -- of the fruit serving a student threw away. We will use this measure to estimate the percentage of fruit servings students wasted.
Fraction of vegetable serving wasted by the student | 30 days
  The tray waste records our researchers collected twice a week (repeated measures) for the duration of the study indicate how much -- 0, one-quarter, one-half, three-quarters, all -- of the vegetable serving a student threw away. We will use this measure to estimate the percentage of vegetable servings students wasted.
Fraction of white milk wasted by the student | 30 days
  The tray waste records our researchers collected twice a week (repeated measures) for the duration of the study indicate how much -- 0, one-quarter, one-half, three-quarters, all -- of the serving of white milk (one pint) a student threw away. We will use this measure to estimate the percentage of white milk servings students wasted.
Fraction of flavored milk wasted by the student | 30 days
  The tray waste records our researchers collected twice a week (repeated measures) for the duration of the study indicate how much -- 0, one-quarter, one-half, three-quarters, all -- of the serving of flavored milk (one pint) a student threw away. We will use this measure to estimate the percentage of flavored milk servings students wasted.
Fraction of entree wasted by the student | 30 days
  The tray waste records our researchers collected twice a week (repeated measures) for the duration of the study indicate how much -- 0, one-quarter, one-half, three-quarters, all -- of the entree serving a student threw away. We will use this measure to estimate the percentage of entree servings students wasted.
Proportion of prepared fruit servings that students took | 75 days
  Cafeterias in the study provided us with food production records that provide daily records of the number of fruit servings cafeteria staff prepared and the number of fruit servings students took. To calculate the proportion of prepared fruit servings taken by students we will divide the number of servings students took by the total number of servings prepared.
Proportion of prepared vegetable servings that students took | 75 days
  Cafeterias in the study provided us with food production records that provide daily records of the number of vegetable servings cafeteria staff prepared and the number of vegetable servings students took. To calculate the proportion of prepared vegetable servings taken by students we will divide the number of servings students took by the total number of servings prepared.
Proportion of prepared entree servings that students took | 75 days
  Cafeterias in the study provided us with food production records that provide daily records of the number of entree servings cafeteria staff prepared and the number of entree servings students took. To calculate the proportion of prepared entree servings taken by students we will divide the number of servings students took by the total number of servings prepared.
Proportion of white milk cartons taken | 75 days
  Cafeterias in the study provided us with food production records that provide daily records of the number of white milk cartons made available and the number of white milk cartons students took. To calculate the proportion of white milk cartons taken by students we will divide the number of servings students took by the total number of servings prepared.
Proportion of flavored milk cartons taken | 75 days
  Cafeterias in the study provided us with food production records that provide daily records of the number of flavored milk cartons made available and the number of flavored milk cartons students took. To calculate the proportion of flavored milk cartons taken by students we will divide the number of servings students took by the total number of servings prepared.
Percentage of total students that took a fruit serving | 75 days
  Cafeterias in the study provided us with food production records that provide daily records of the number of fruit servings prepared and the total number of students who received a school lunch. To calculate the percentage of students who took a fruit serving we will divide the number of servings students took by the total number of students who received lunch.
Percentage of total students that took a vegetable serving | 75 days
  Cafeterias in the study provided us with food production records that provide daily records of the number of vegetable servings prepared and the total number of students who received a school lunch. To calculate the percentage of students who took a vegetable serving we will divide the number of servings students took by the total number of students who received lunch.
Percentage of total students that took an entree serving | 75 days
  Cafeterias in the study provided us with food production records that provide daily records of the number of entree servings prepared and the total number of students who received a school lunch. To calculate the percentage of students who took an entree serving we will divide the number of servings students took by the total number of students who received lunch.
Percentage of total students that took a carton of white milk | 75 days
  Cafeterias in the study provided us with food production records that provide daily records of the number of white milk cartons made available the total number of students who received a school lunch. To calculate the percentage of students who took a carton of white milk we will divide the number of servings students took by the total number of students who received lunch.
Percentage of total students that took a carton of flavored milk | 75 days
  Cafeterias in the study provided us with food production records that provide daily records of the number of flavored milk cartons made available the total number of students who received a school lunch. To calculate the percentage of students who took a carton of flavored milk we will divide the number of servings students took by the total number of students who received lunch.
Percentage of fidelity assessments that returned positive marks | 36 days
  Throughout the study, researchers conducted fidelity assessments to make sure the schools maintained the interventions. These process control measures are the ratio of successful fidelity checks to the total number. Researchers conducted these assessments during each day they collected tray waste measures and during a randomly selected non-tray waste collection date once a month.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Hanks, PhD, Principal Investigator — Ohio State University; Haleigh Gaines, MS,RD, Study Director — Ohio State University
Locations (6):
- United States (6):
  - Champion Middle School, Columbus, Ohio
  - Hilltonia Middle School, Columbus, Ohio
  - Buckeye Middle School, Columbus, Ohio
  - Mifflin Middle School, Columbus, Ohio
  - Medina Middle School, Columbus, Ohio
  - Johnson Park Middle School, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
We agree to share the study data with researchers who request access. While we will not publicly post the data, we will provide them through an electronic link. None of the data contain unique identifiers.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data are available as of October 29, 2019 and will be available until December 31, 2020.
Access Criteria: Those interested in acquiring the data can contact Dr. Andrew Hanks at hanks.46@osu.edu.